CLINICAL TRIAL: NCT06138379
Title: The Effect of Video-Assisted Education Given to Patients With Liver Transplantation in the Line of Health Belief Model on Adaptation to Disease and Drug Use
Brief Title: Video-supported Training in Line With the Health Belief Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Associate Professor Dr. Zeliha CENGİZ, Head of the Department of Nursing Principles, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/4674
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Education

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a randomized controlled experimental study. The population of the research will consist of adult patients who received liver transplantation at İnönü University Turgut Özal Medical Center. The sample will consist of 90 patients determined by power analysis.
Masking Description: It will be collected using the Patient Introduction Form, Chronic Disease Adaptation Scale, Immunosuppressive Drug Use Compliance Scale and Rational Drug Use Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No Intervention: Control group The research will begin after obtaining the necessary legal and ethical permissions to collect data. At this stage of the research, participants who agree to participate in the research will be asked to fill out an informed consent form. All forms will be filled in to obtain pre-test data for the research.
  These individuals who receive and continue to receive standard care will be informed about the research. Pre-test and post-test data from the control group will be obtained simultaneously with the study groups.
- 1. Experimental Group (Experimental): Experimental: Experimental group given video-supported training in line with the health belief model.
  All forms (Patient Information Monitoring Form, Chronic Disease Adaptation Scale, Rational Drug Use Scale and Immunosuppressive Drug Form Scale) will be filled in to obtain pre-test data for the research. Individuals will be trained according to the training materials prepared for the Health Belief Model. They will be monitored one day each week. After 30 days, all forms will be filled out again to examine the sustainability of the training data.
  Interventions: Other: Experimental: 1st Experimental Group
- 2. Experimental Group (Experimental): Experimental: The experimental group was given video-supported training in line with Classical Education.
  All forms (Patient Information Monitoring Form, Chronic Disease Adaptation Scale, Rational Drug Use Scale and Immunosuppressive Drug Form Scale) will be filled in to obtain pre-test data for the research. Individuals will be trained according to the training materials prepared for the Health Belief Model. They will be monitored one day each week. After 30 days, all forms will be filled out again to examine the sustainability of the training data.
  Interventions: Other: Experimental: 2nd Experimental Group

INTERVENTIONS:
Other: Experimental: 1st Experimental Group — Individuals will be sent relevant educational videos after liver transplantation and asked to watch them.
  Other Names: Video-supported teaching in line with the Health Belief Model
  Arms: 1. Experimental Group
Other: Experimental: 2nd Experimental Group — Individuals will be sent relevant educational videos after liver transplantation and asked to watch them.
  Other Names: Video assisted teaching
  Arms: 2. Experimental Group

SUMMARY:
Summary The only treatment method for those with incurable, irreversible, progressive, acute or chronic liver disease is liver transplantation. Compliance with the disease and immunosuppressive treatment has an important place in the success of transplants. This study was planned to examine the effect of video-supported education given to liver transplant patients in line with the Health Belief Model on adaptation to chronic disease and medication use.

The research will be conducted as a randomized controlled experimental study. The population of the research will consist of adult patients who received liver transplantation at İnönü University Turgut Özal Medical Center. The sample will consist of 90 patients determined by power analysis. Patients will be divided into three groups: control (n=30), 1st experiment (n=30) and 2nd experiment (n=30). Data will be collected between August 2023 and December 2023 using the Patient Information Form, Chronic Disease Adaptation Scale, Immunosuppressive Drug Use Compliance Scale and Rational Drug Use Scale. Video-supported training will be provided to patients in the experimental group to increase compliance with the disease and immunosuppressive treatment and to ensure rational drug use. Patients in the 1st experimental group will receive video-supported training in line with the Health Belief Model for one month, and patients in the 2nd experimental group will receive video-supported standard training for one month. This video training will be given to the experimental group patients outside the routine nursing care of the clinic. The video-supported training is planned to last 20-30 minutes. Nursing care in the routine practice of the clinic will be applied to the control group. Evaluation of data; It will be done with number, percentage, mean, standard deviation, chi-square, paired t test, t test analysis in independent groups, ANOVA and ANCOVA.

As a result, it is predicted that video-supported education will increase compliance with chronic disease and medication use and reduce post-transplant symptoms and discomfort caused by these symptoms.

DETAILED DESCRIPTION:
Although there are studies on video-supported education in the literature, no research has been found examining the effect of video-assisted education in line with SIM on disease adaptation and medication use in liver transplant patients. For this reason, in this research, it is aimed to minimize the risks by obtaining information about the beliefs and tendencies of the patients, adapting to chronic diseases and medication use, with the video-supported training prepared in line with the use of SIM as an effective tool. The research is unique because it is the first study comparing the education provided with SIM and standard education. When the difference between the training given with SIM and standard training is determined, it can be stated with strong evidence that compliance with the disease and medication may be due to the training given with the model.

ELIGIBILITY:
Inclusion Criteria:• No communication problems,

* Those who are 18 years of age and over,
* At least 2 months and at most 2 years have passed since the transplant,
* Having a device (phone, tablet, computer, etc.) that can watch the video,
* Patients who are literate will be included in the study.

Exclusion Criteria:• Do not watch research videos,

* Communication problems occur,
* Patients with distressing medical conditions will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Patient Introduction Form | 6 months
  It is a form prepared by the researcher and examines the sociodemographic and medical characteristics of liver transplant patients. This form includes 11 questions to determine the patients' age, gender, marital status, education level, employment status, income level, how long they have had liver disease, additional diseases, the presence of people assisting in the care, how long ago the transplant was performed, and the donor type.
Chronic Illness Adjustment Scale | 6 months
  It was developed by Derya Atik and Hilal Karatepe in 2016. The scale consists of 25 items. It consists of three subscales: Physical Adaptation (11 items), Social Adaptation (7 items), and Psychological Adaptation (7 items). Subdimensions of the scale; 1. Physical Harmony; Items 1, 9, 10, 13, 14, 15, 16, 18, 22, 23, 24 (minimum 11, maximum 55 points), 2. Social Cohesion; 2nd, 3rd, 5th, 7th, 17th, 19th, 25th items (minimum 7, maximum 35 points), 3. Psychological Adjustment; Items 4, 6, 8, 11, 12, 20, 21 measure (minimum 7, maximum 35 points). Scoring: 1st, 2nd, 3rd, 4th, 7th, 8th, 9th, 10th, 11th, 13th, 14th, 15th, 16th, 18th, 21st, 22nd, The 23rd items are normal (in the form of 1,2,3,4,5), the 5th, 6th, 12th, 17th, 19th, 20th, 24th, 25th items are reverse (5,4,3,2). It is scored as .1). The total score that can be obtained from the scale is 125. Higher scores from the subscales and/or the entire scale mean that patients' adaptation levels to the disease increase.
Compliance with Immunosuppressive Medication Use Scale | 6 months
  In the scale developed by Özdemir, the compliance with medication use of patients who have had solid organ transplants and are taking immunosuppressive drugs is evaluated. In order for the scale to be applied, patients must complete at least two months after transplantation. The scale consists of 11 items in total. Scoring is done with a 5-point and 2-point Likert type rating. The scale includes positive and negative expressions. Positive statements are 4 and 6, and negative statements are 1, 2, 3, 5, 7, 8, 9, 10 and 11. Positive statements are scored from 1 to 5, while negative statements are scored from 5 to 1. For positive items, 1 point is given for a 'yes' answer and 5 points are given for a 'no' answer. The lowest score of the scale is 11 and the highest score is 55. As the score from the scale increases, compliance with medication use increases, and as the score decreases, compliance with medication use decreases. Cronbach's alpha value was calculated as 0.611 by Özdemir.
Rational Drug Use Scale | 6 months
  It consists of 21 items and a single dimension. Items are scored on a 5-point Likert-type scale according to the situations in which they realize the statements (1-Never, 2-Rarely, 3-Occasionally, 4-Often and 5-Always). Only the 17th item in the scale is reverse scored. After the reverse-scored item is translated, the sum of all scale items gives the "total scale score". The total score of AİKÖ varies between 21 and 105. As the total score obtained from ADAS increases, rational drug use increases. When evaluating the total score received from AİKÖ; If the total score is between 21 and 52, it is scored as low, between 53 and 67, as medium, and between 68 and 105, it is scored as high.

CONTACTS AND LOCATIONS:
Overall Officials: Sezai Yılmaz, Prof Dr, Study Director — Turgut Ozal Medical Center
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can be used as a source for other research.